CLINICAL TRIAL: NCT04834232
Title: Comparative Study Between Iliac Vein Stenting and Compression Therapy in Recurrent Venous Ulceration
Brief Title: Iliac Vein Stenting and Compression Therapy in Recurrent Venous Ulceration
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed hesham abdelrahem husiein, principal investigator, Assiut University
Other Study IDs: stenting & compression therapy
Record Dates: First submitted 2020-09-26; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Venous Ulcer Recurrent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: compression therapy — compression bandaging or graduated compression hosiery consists of applying a type of elastic device, mainly on the limbs, to exert a controlled pressure on the lower limbs. The controlled pressure exerted by medical compression stockings reduces the diameter of major veins, thereby increasing the velocity and volume of blood flow, along with conditions beneficial for the healing of chronic inflammatory disorders (e.g. cellulitis, erysipelas, venous leg ulcers, etc.), through reduced pro-inflammatory cytokine levels and higher levels of the anti-inflammatory cytokines.
Procedure: iliac vein stenting — using x-ray guidance (fluoroscopy) to place a an expandable metal mesh tube against the vein walls, acting as a scaffold to keep the veins open and improve blood flow

SUMMARY:
Comparing the result of of iliac vein stenting and compression therapy in management of recurrent venous ulceration.

DETAILED DESCRIPTION:
Venous ulceration is the most common etiology of lower extremity ulceration, approximately affecting almost 1% of the world's population. although its overall prevalence is relatively low, the refractory nature of venous ulceration increases morbidity, mortality , the patient's quality of life, and have a significant financial burden on the global budget. the primary risk factors are: old age, obesity deep venous thrombosis, phlebitis and previous leg injuries.

Iliac vein compression is a prevalent finding in patients with venous system pathology. It has a variety of causes, including May-Turner syndrome, endometriosis, bladder distension, common iliac artery aneurysm or internal iliac artery aneurysm.

venous compression becomes clinically significant when there's an increase in venous pressure, which in turn causes venous insufficiency. This contributes to the development of a state of chronic venous stasis, which sequentially causes pooling of blood, triggers further capillary damage and activates inflammatory mediators with the end result of venous ulcer development and impaired wound healing.

Located on bony prominences, venous ulcers are typically shallow, irregular with granulation tissue and fibrin present in their bases. A careful physical examination is required for a proper diagnosis, but he clinical challenge remains in its management, which includes prevention or the treatment of the clinical implications.

Treatment modalities should always be directed to the cause of the ulcer; they can be divided into:

* non invasive management, such as medical therapy, bandaging and dressings.
* invasive, such as endovascular and surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* iliac vein compression.
* competent superficial venous system.
* isolated iliac vein lesion.
* patent femoropopliteal segment.
* ulcers located in the gaiter area.
* age > 12 years
* patients with ulcers located in the gaiter area, along with the following associated symptoms: leg heaviness, pain, varicose veins, edema, hemosedrin staining, pruritus, venous dermatitis, lipodermatoscelrosis, telangiectasias, corona phlebectatica, atrophie blanche and deformity of the leg.

Exclusion Criteria:

* patients with arterial disease in the same limb.
* patients with history of phlebitis.
* patients with congenital venous malformation
* patients with malignancy.
* patients with raised renal chemistry.
* patients with skin allergy.
* diabetic neuropathic ulcer.
* atypical site of venous ulcer.
* acute onset DVT.
* age < 12 years.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients fulfilling both the inclusion and the exclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
ulcer healing within 6 months | baseline
  comparing the results of both modalities in recurrent venous ulcer healing

SECONDARY OUTCOMES:
patency on stents | baseline
  primary assisted patency included those requiring reintervention to maintain patency; and secondary patency was defined as stents that were blocked and successfully reopened.
compliance | baseline
  to anticoagulation in case of stenting, or to elastic stocking in case of compression therapy, using methods that include patient self-reporting and clinical estimates
assessment of venous disability score (VDS) | baseline
  the VDS evaluates the effect of venous disease by quantifying the level of work based disability.
  It is scored on a scale of 0 to 3 (with 0 being the least severe and 3 the most severe), based on the ability to work an 8-hour day with or without provisions for external support.
assessment of venous clinical severity score | baseline
  the score is obtained by imaging vein segments with duplex Doppler or phlebography.
  It includes 9 hallmarks of venous disease, each scored on a severity scale from 0 to 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

REFERENCES:
- [Background] Raju S. Best management options for chronic iliac vein stenosis and occlusion. J Vasc Surg. 2013 Apr;57(4):1163-9. doi: 10.1016/j.jvs.2012.11.084. Epub 2013 Feb 20. PMID 23433816
- [Background] Xie T, Ye J, Rerkasem K, Mani R. The venous ulcer continues to be a clinical challenge: an update. Burns Trauma. 2018 Jun 15;6:18. doi: 10.1186/s41038-018-0119-y. eCollection 2018. PMID 29942813
- [Background] George R, Verma H, Ram B, Tripathi R. The effect of deep venous stenting on healing of lower limb venous ulcers. Eur J Vasc Endovasc Surg. 2014 Sep;48(3):330-6. doi: 10.1016/j.ejvs.2014.04.031. Epub 2014 Jun 18. PMID 24953000
- [Background] Nair B. Compression therapy for venous leg ulcers. Indian Dermatol Online J. 2014 Jul;5(3):378-82. doi: 10.4103/2229-5178.137822. No abstract available. PMID 25165679